CLINICAL TRIAL: NCT00550173
Title: A Randomized Phase 2 Study Comparing Erlotinib-Pemetrexed, Pemetrexed Alone, and Erlotinib Alone, as Second-Line Treatment for Non-Smoker Patients With Locally Advanced or Metastatic Nonsquamous Non-Small Cell Lung Cancer
Brief Title: A Study for Non-Smoker Patients With Nonsquamous Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10725; H3E-MC-S103 (Other: Eli Lilly and Company)
Record Dates: First submitted 2007-10-25; First posted 2007-10-29 (Estimated); Results first posted 2013-02-13 (Estimated); Last update posted 2013-02-13 (Estimated); Status verified 2013-01

CONDITIONS: Non-Small-Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Pemetrexed + Erlotinib (Experimental): Pemetrexed 500 milligrams per meter squared (mg/m^2) of body surface area, administered by intravenous (IV) infusion on Day 1 plus erlotinib 150 mg orally once daily on Day 2 through Day 14 of each 21-day cycle until disease progression or unacceptable toxicity developed or up to 38 months.
  Interventions: Drug: pemetrexed; Drug: erlotinib
- Erlotinib (Active Comparator): Erlotinib 150 mg, administered orally once daily in each 21-day cycle until disease progression or unacceptable toxicity developed or up to 38 months.
  Interventions: Drug: erlotinib
- Pemetrexed (Active Comparator): Pemetrexed 500 mg/m^2 of body surface area, administered by IV infusion on Day 1 of each 21-day cycle until progression or unacceptable toxicity developed or up to 38 months.
  Interventions: Drug: pemetrexed

INTERVENTIONS:
Drug: pemetrexed — 500 milligrams per meter squared (mg/m^2), intravenous (IV), every (q) 21 days until progression or unacceptable toxicity develops
  Other Names: LY231514; Alimta
  Arms: Pemetrexed; Pemetrexed + Erlotinib
Drug: erlotinib — 150 mg, orally, once daily until progression or unacceptable toxicity develops
  Arms: Erlotinib; Pemetrexed + Erlotinib

SUMMARY:
The purpose of this study is to compare the combination of erlotinib and pemetrexed versus either pemetrexed alone and erlotinib alone, in terms of progression-free survival (time until the objective worsening of the disease) in patients who have never smoked and have locally advanced or metastatic Nonsquamous Non-Small Cell Lung Cancer who have failed a first-line chemotherapy treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with locally advanced or metastatic nonsquamous non-small cell lung cancer
* Patients must be non-smokers
* Patients must have at least one measurable lesion
* Performance status of 0 to 2 on the Eastern Cooperative Oncology Group Scale
* Patients must have failed only one prior chemotherapy regimen and must be considered eligible for further chemotherapy following progression of their disease.

Exclusion Criteria:

* Patients who have received treatment within the last 30 days with a drug that has not received regulatory approval for any indication
* Patients who have previously received treatment with drugs against the human epidermal growth factor receptors
* Patients who have previously received treatment with drugs which have similar targets as Pemetrexed
* Patients who have any known significant ophthalmologic abnormalities of the surface of the eye
* Patients who have a history of severe hypersensitivity reaction to erlotinib or pemetrexed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 247 (Actual)
Dates: Start 2007-11; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (29):
- Brazil (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barretos
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ijuí
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., São Paulo
- China (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beijing
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nanning
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shanghai
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shatin, Hong Kong
- India (11):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ahmedabad
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bhopal
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyderabaad
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jaipur
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kochi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kolkata
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madurai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mohali
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mumbai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New Delhi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Visakhapatnam
- South Korea (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jinju
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Suwon
- Taiwan (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Changhua
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taichung
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taoyuan District
- United Kingdom (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Poole, Dorset
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chelmsford, Essex
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aberdeen, Scotland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guildford, Surrey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Manchester, United Kingdom

REFERENCES:
- [Derived] Lee DH, Lee JS, Kim SW, Rodrigues-Pereira J, Han B, Song XQ, Wang J, Kim HK, Sahoo TP, Digumarti R, Wang X, Altug S, Orlando M. Three-arm randomised controlled phase 2 study comparing pemetrexed and erlotinib to either pemetrexed or erlotinib alone as second-line treatment for never-smokers with non-squamous non-small cell lung cancer. Eur J Cancer. 2013 Oct;49(15):3111-21. doi: 10.1016/j.ejca.2013.06.035. Epub 2013 Jul 24. PMID 23890768
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pemetrexed + Erlotinib | Erlotinib | Pemetrexed
Started | 81 | 82 | 84
Qualified Participants | 78 (Participants with tumors of nonsquamous histology) | 82 (Participants with tumors of nonsquamous histology) | 80 (Participants with tumors of nonsquamous histology)
Not Discontinued at 18 Months | 9 | 19 | 11
Completed | 9 | 19 | 11
Not Completed | 72 | 63 | 73
Not completed — Death | 45 | 38 | 50
Not completed — Physician Decision | 1 | 2 | 2
Not completed — Withdrawal by Subject | 9 | 12 | 17
Not completed — Sponsor Decision | 13 | 7 | 1
Not completed — Lost to Follow-up | 4 | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Pemetrexed + Erlotinib: Pemetrexed 500 mg/m^2 of body surface area, administered by IV infusion on Day 1 plus erlotinib 150 mg orally once daily on Day 2 through Day 14 of each 21-day cycle until disease progression or unacceptable toxicity developed or up to 38 months.
- Total: Total of all reporting groups
Arm/Group | Pemetrexed + Erlotinib | Erlotinib | Pemetrexed | Total
Number analyzed (Participants) | 78 | 82 | 80 | 240
Age Continuous [Mean (Standard Deviation); unit: years] | 56.0 (11.72) | 53.9 (10.49) | 56.1 (13.04) | 55.3 (11.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 54 | 45 | 157
  Male | 20 | 28 | 35 | 83
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 18 | 6 | 11 | 35
  African | 2 | 0 | 1 | 3
  East Asian (enrolled in an East Asian country) | 41 | 49 | 43 | 133
  East Asian (enrolled in non-East Asian Country) | 4 | 2 | 1 | 7
  West Asian | 13 | 25 | 24 | 62
Region of Enrollment [Number; unit: participants]
  Australia | 3 | 0 | 0 | 3
  Brazil | 15 | 5 | 8 | 28
  China | 14 | 17 | 15 | 46
  Hong Kong | 0 | 3 | 2 | 5
  India | 15 | 27 | 25 | 67
  Korea, Republic of | 20 | 20 | 13 | 53
  Taiwan | 7 | 9 | 13 | 29
  United Kingdom | 4 | 1 | 4 | 9
Height at Baseline [Mean (Standard Deviation); unit: centimeter (cm)] | 159.3 (8.70) | 160.3 (8.38) | 160.1 (8.84) | 159.9 (8.61)
Weight at Baseline [Mean (Standard Deviation); unit: kilogram (kg)] | 59.6 (11.76) | 59.9 (12.17) | 58.9 (10.82) | 59.5 (11.56)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per meter squared (kg/m^2)] — BMI is an estimate of body fat based on body weight divided by height squared.
  kilogram per meter squared (kg/m^2) | 23.5 (4.54) | 23.3 (3.87) | 23.0 (3.87) | 23.2 (4.09)
Body Surface Area (BSA) [Mean (Standard Deviation); unit: meter squared (m^2)] | 1.6 (0.17) | 1.6 (0.18) | 1.6 (0.17) | 1.6 (0.17)
Eastern Cooperative Oncology Group Performance Status (ECOG PS) [Number; unit: participant] — ECOG PS Scale: 0 = fully active, able to perform all pre-disease activities unrestricted; 1 = restricted in physically strenuous activity but ambulatory, able to carry out light or sedentary activities; 2 = ambulatory, capable of all self-care but unable to carry out any work activities, up and about more than 50% of waking hours; 3 = capable of only limited self-care, confined to bed or chair more than 50% of waking hours; 4 = completely disabled, cannot carry on any self-care, totally confined to bed or chair; 5 = Dead.
  participant
    0 | 10 | 20 | 16 | 46
    1 | 61 | 56 | 60 | 177
    2 | 6 | 6 | 4 | 16
    3 | 1 | 0 | 0 | 1
Histological Subtype [Number; unit: participants]
  Adenocarcinoma (adeno) | 72 | 76 | 77 | 225
  Non-adenocarcinoma (non-adeno) | 6 | 6 | 3 | 15

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: PFS is defined as the time from randomization to the first date of progressive disease (PD; either objectively determined or clinical progression) or death from any cause. PD was defined as at least a 20% increase in sum of longest diameter of target lesions as assessed by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.0 guidelines. Time to disease progression was censored at the date of death.
Time Frame: Randomization to measured PD up to 38 months
Population: Qualified Intent to Treat (Q-ITT) Population defined as all participants with nonsquamous histology, who were randomized to therapy.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Pemetrexed + Erlotinib: Pemetrexed 500 mg/m^2 of BSA, administered by IV infusion on Day 1 plus erlotinib 150 mg orally once daily on Day 2 through Day 14 of each 21-day cycle until disease progression or unacceptable toxicity developed or up to 38 months.
- Pemetrexed: Pemetrexed 500 mg/m^2 of BSA, administered by IV infusion on Day 1 of each 21-day cycle until progression or unacceptable toxicity developed or up to 38 months.
Arm/Group | Pemetrexed + Erlotinib | Erlotinib | Pemetrexed
Number analyzed (Participants) | 78 | 82 | 80
months | 7.4 [4.4 to 12.9] | 3.8 [2.7 to 6.3] | 4.4 [3.0 to 6.0]
Statistical Analysis 1: Comparison: Pemetrexed + Erlotinib vs Erlotinib vs Pemetrexed; Overall; Global null hypothesis was rejected at 2-sided 0.2 significance level; Test type: Superiority or Other; p = 0.003, Regression, Cox — If global test across 3 arms is significant at a 2-sided 0.2 level, then conduct 2-sided pairwise tests between combination and each single agent under the global model. Significance is claimed only if both the global and pairwise tests p<0.05; Model is adjusted to covariates ECOG PS (0/1 vs.2), histological subtype (adeno vs. non-adeno), race (East Asian and non-East Asian) and gender
Statistical Analysis 2: Comparison: Pemetrexed + Erlotinib vs Erlotinib; Primary Analysis; Global null hypothesis was rejected at 2-sided 0.2 significance level; Test type: Superiority or Other; p = 0.002, Regression, Cox — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.57, 95% CI 2-sided [0.40 to 0.81]
Statistical Analysis 3: Comparison: Pemetrexed + Erlotinib vs Pemetrexed; Primary Analysis; Global null hypothesis was rejected at 2-sided 0.2 significance level; Test type: Superiority or Other; p = 0.005, Regression, Cox — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.58, 95% CI 2-sided [0.39 to 0.85]
Statistical Analysis 4: Comparison: Erlotinib vs Pemetrexed; Secondary Analysis; Global null hypothesis was rejected at 2-sided 0.2 significance level; Test type: Superiority or Other; p = 0.959, Regression, Cox — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Hazard Ratio, log = 0.99, 95% CI 2-sided [0.70 to 1.40]

2. Secondary Outcome: Percentage of Participants With a Tumor Response of Complete Response (CR) or Partial Response (PR) [Tumor Response Rate (TRR)]
Description: TRR was defined as the number of responders (complete or partial) divided by the number of participants qualified for tumor response, as assessed using the RECIST version 1.0 guideline, multiplied by 100. RECIST guidelines: CR was defined as the disappearance of all target and non-target lesions and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 millimeter (mm) and normalization of tumor marker level of non-target lesions; PR was defined as at least a 30% decrease in sum of longest diameter of target lesions.
Time Frame: Randomization to measured disease progression up to 38 months
Population: Q-ITT Population - Tumor Analyzable (Q-ITT-TA) Population: defined as all participants with nonsquamous histology, who were randomized to therapy and had measurable or evaluable lesions at baseline.
Measure: Number; unit: percentage of participants
Arm/Group | Pemetrexed + Erlotinib | Erlotinib | Pemetrexed
Number analyzed (Participants) | 76 | 82 | 80
percentage of participants | 44.7 | 29.3 | 10.0
Statistical Analysis 1: Comparison: Pemetrexed + Erlotinib vs Erlotinib vs Pemetrexed; Test type: Superiority or Other; p < 0.001, Regression, Logistic; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Pemetrexed + Erlotinib vs Erlotinib; Test type: Superiority or Other; p = 0.031, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 2.09, 95% CI 2-sided [1.07 to 4.09]
Statistical Analysis 3: Comparison: Pemetrexed + Erlotinib vs Pemetrexed; Test type: Superiority or Other; p < 0.001, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 7.68, 95% CI 2-sided [3.19 to 18.48]
Statistical Analysis 4: Comparison: Erlotinib vs Pemetrexed; Test type: Superiority or Other; p = 0.004, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio, log = 0.27, 95% CI 2-sided [0.11 to 0.66]

3. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from randomization to the date of death from any cause.
Time Frame: Baseline to date of death from any cause up to 45.5 months
Population: Q-ITT Population: defined as all participants with nonsquamous histology, who were randomized to therapy. Survival time was censored at the date of last contact for participants who were still alive or lost to follow-up, number of participants censored 35 (pemetrexed plus erlotinib), 44 (erlotinib) and 31 (pemetrexed).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed + Erlotinib | Erlotinib | Pemetrexed
Number analyzed (Participants) | 78 | 82 | 80
months | 20.5 [17.1 to 25.0] | 22.8 [18.2 to 29.5] | 17.7 [11.8 to 25.3]
Statistical Analysis 1: Comparison: Pemetrexed + Erlotinib vs Erlotinib vs Pemetrexed; Test type: Superiority or Other; p = 0.194, Regression, Cox; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Pemetrexed + Erlotinib vs Erlotinib; Test type: Superiority or Other; p = 0.747, Regression, Cox; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.08, 95% CI 2-sided [0.69 to 1.67]
Statistical Analysis 3: Comparison: Pemetrexed + Erlotinib vs Pemetrexed; Test type: Superiority or Other; p = 0.168, Regression, Cox; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.49 to 1.13]
Statistical Analysis 4: Comparison: Erlotinib vs Pemetrexed; Test type: Superiority or Other; p = 0.094, Regression, Cox; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.44, 95% CI 2-sided [0.94 to 2.21]

4. Secondary Outcome: Number of Participants With Adverse Events
Description: A summary of serious and all other non-serious adverse events (AEs), which include AEs reported for pharmacological toxicity, is located in the Reported Adverse Event module.
Time Frame: Randomization up to 39 months
Population: Safety Population defined as non-squamous participants who received at least 1 dose of study therapy (pemetrexed plus erlotinib or pemetrexed or erlotinib). One participant was assigned to pemetrexed (single therapy) but received erlotinib (single therapy) at first cycle and this lead to the discrepancy of participants for the safety analysis.
Measure: Number; unit: participants
Arm/Group | Pemetrexed + Erlotinib | Erlotinib | Pemetrexed
Number analyzed (Participants) | 78 | 83 | 80
participants
  Serious Adverse Events | 25 | 18 | 22
  Other Non-Serious Adverse Events | 72 | 76 | 67

5. Secondary Outcome: Percentage of Participants With CR, PR, and Stable Disease (SD) - Disease Control Rate (DCR)
Description: DCR was defined as the percentage of participants with CR, PR, or SD divided by the number of randomized and treated participants as assessed using the RECIST criteria. CR was defined as the disappearance of all target lesions; PR was defined as 1) at least a 30% decrease in sum of longest diameter of target lesions or 2) complete disappearance of target lesions, with persistence (but not worsening) of 1 or more non-target lesions; PD was defined as at least a 20% increase in sum of longest diameter of target lesions; SD was defined as small changes that did not meet the above criteria.
Time Frame: Randomization to disease progression up to 38 months
Population: Q-ITT-TA Population: defined as all participants, with nonsquamous histology, who were randomized to therapy and had measurable or evaluable lesions at baseline.
Measure: Number; unit: percentage of participants
Arm/Group | Pemetrexed + Erlotinib | Erlotinib | Pemetrexed
Number analyzed (Participants) | 76 | 82 | 80
percentage of participants | 64.5 | 52.4 | 56.3
Statistical Analysis 1: Comparison: Pemetrexed + Erlotinib vs Erlotinib vs Pemetrexed; Test type: Superiority or Other; p = 0.306, Regression, Logistic; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Pemetrexed + Erlotinib vs Erlotinib; Test type: Superiority or Other; p = 0.127, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.66, 95% CI 2-sided [0.87 to 3.18]
Statistical Analysis 3: Comparison: Pemetrexed + Erlotinib vs Pemetrexed; Test type: Superiority or Other; p = 0.318, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.40, 95% CI 2-sided [0.72 to 2.71]
Statistical Analysis 4: Comparison: Erlotinib vs Pemetrexed; Test type: Superiority or Other; p = 0.599, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.18, 95% CI 2-sided [0.63 to 2.22]

6. Secondary Outcome: Time to Worsening of Symptoms (TWS) on Lung Cancer Symptoms Scale (LCSS)
Description: TWS assessed using the LCSS a participant rated lung cancer instrument which consisted of 9 disease related symptoms and quality of life (QoL) items, with 6 subscales related to major lung cancer symptoms (appetite, cough, fatigue, dyspnea, hemoptysis, and pain) and 3 summation items related to QoL (activity status, symptomatic distress, and overall QoL). Each item is marked on a visual analog scale (VAS) 0 (low symptoms/QoL items) to 100 (high symptoms/QoL items). The mean of the 6 subscales is used to calculate the average symptom burden index. TWS was measured from the date of study enrollment to the first date of a worsening in any 1 of the 6 LCSS symptom-specific items (as defined by a VAS 15-mm increase from baseline in the patient-reported score for any of these 6 items).
Time Frame: Randomization to first date of worsening of any of 6 LCSS symptom specific items or up to 12.4 months
Population: A subset of the Q-ITT Population that included participants with LCSS results; Q-ITT Population: defined as all participants, with nonsquamous histology, who were randomized to therapy.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed + Erlotinib | Erlotinib | Pemetrexed
Number analyzed (Participants) | 70 | 71 | 65
months | 1.0 [0.9 to 1.6] | 0.8 [0.8 to 1.2] | 1.5 [1.0 to 2.1]
Statistical Analysis 1: Comparison: Pemetrexed + Erlotinib vs Erlotinib vs Pemetrexed; Test type: Superiority or Other; p = 0.013, Regression, Cox; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Pemetrexed + Erlotinib vs Erlotinib; Test type: Superiority or Other; p = 0.007, Regression, Cox — Model is adjusted to covariates ECOG PS (0/1 vs.2), histological subtype (adeno vs. non-adeno), race (East Asian and non-East Asian) and gender; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.59, 95% CI 2-sided [0.41 to 0.87]
Statistical Analysis 3: Comparison: Pemetrexed + Erlotinib vs Pemetrexed; Test type: Superiority or Other; p = 0.700, Regression, Cox; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.62 to 1.38]
Statistical Analysis 4: Comparison: Erlotinib vs Pemetrexed; Test type: Superiority or Other; p = 0.023, Regression, Cox; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.64, 95% CI 2-sided [0.44 to 0.94]

7. Secondary Outcome: Number of Participants With Mutated or Non-Mutated Epidermal Growth Factor Receptor (EGFR) Genotype Status
Description: EGFR mutation status was defined as: participants with any mutations detected were categorized as mutated and participants without any mutations detected were categorized as non-mutated.
Time Frame: Randomization to date of PD or death up to 38 months
Population: A subset of the Q-ITT Population who had EGFR samples; Q-ITT Population: defined as all participants with nonsquamous histology, who were randomized to therapy.
Measure: Number; unit: participants
Arm/Group | Pemetrexed + Erlotinib | Erlotinib | Pemetrexed
Number analyzed (Participants) | 22 | 16 | 15
participants
  Mutated | 7 [lower limit 7.1] | 8 | 9
  Non-mutated | 10 | 6 | 3
  Mutation status unknown (treated as missing) | 5 | 2 | 3
Statistical Analysis 1: Comparison: Pemetrexed + Erlotinib vs Erlotinib vs Pemetrexed; Test type: Superiority or Other; p = 0.040, Regression, Cox
Statistical Analysis 2: Comparison: Pemetrexed + Erlotinib vs Erlotinib; Test type: Superiority or Other; p = 0.241, Regression, Cox; Hazard Ratio (HR) = 0.62, 95% CI 2-sided [0.27 to 1.38]
Statistical Analysis 3: Comparison: Pemetrexed + Erlotinib vs Pemetrexed; Test type: Superiority or Other; p = 0.011, Regression, Cox; Hazard Ratio (HR) = 0.32, 95% CI 2-sided [0.14 to 0.78]
Statistical Analysis 4: Comparison: Erlotinib vs Pemetrexed; Test type: Superiority or Other; p = 0.128, Regression, Cox; Hazard Ratio (HR) = 1.90, 95% CI 2-sided [0.83 to 4.36]

8. Secondary Outcome: Probability of OS at 12 Months
Description: OS time is censored at the date of last contact for participants who were still alive or lost to follow-up.
Time Frame: Month 12
Population: Q-ITT Population: defined as all participants with nonsquamous histology, who were randomized to therapy.
Measure: Number (95% Confidence Interval); unit: percent chance of survival
Arm/Group | Pemetrexed + Erlotinib | Erlotinib | Pemetrexed
Number analyzed (Participants) | 78 | 82 | 80
percent chance of survival | 40.2 [28.3 to 51.8] | 26.2 [17.2 to 36.1] | 18.1 [9.1 to 29.4]

ADVERSE EVENTS:
Description: One participant was assigned to Pemetrexed (single therapy) but received Erlotinib (single therapy) at the first cycle, this leads to the discrepancy of participants for the safety analysis.
Groups:
- Pemetrexed + Erlotinib: Participants received pemetrexed 500 milligrams per meter squared (mg/m^2) of body surface area, administered by intravenous (IV) infusion on Day 1 plus erlotinib 150 mg orally once daily on Day 2 through Day 14 of each 21 day cycle until disease progression or unacceptable toxicity developed up to 39 months.
- Erlotinib: Participants received erlotinib 150 mg, administered orally once daily in each 21 day cycle until disease progression or unacceptable toxicity developed up to 39 months.
- Pemetrexed: Participants received pemetrexed 500 mg/m^2 of body surface area, administered by intravenous (IV) infusion on Day 1 of each 21 day cycle until progression or unacceptable toxicity developed up to 39 months.
Arm/Group | Pemetrexed + Erlotinib | Erlotinib | Pemetrexed
Serious Adverse Events (participants affected / at risk) | 25/78 | 18/83 | 22/80
Other Adverse Events (participants affected / at risk) | 72/78 | 76/83 | 67/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed + Erlotinib (N=78) | Erlotinib (N=83) | Pemetrexed (N=80)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 0 (0) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Asthenia (General disorders) | 2 (3) | 2 (2) | 1 (1)
Death (General disorders) | 0 (0) | 0 (0) | 1 (1)
Irritability (General disorders) | 0 (0) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 2 (2) | 1 (1)
Sudden death (General disorders) | 0 (0) | 1 (1) | 1 (1)
Hepatitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 3 (4) | 0 (0)
Respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hemiplegia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Nervous system disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Neurotoxicity (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Radicular pain (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Renal failure chronic (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (6) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed + Erlotinib (N=78) | Erlotinib (N=83) | Pemetrexed (N=80)
Anaemia (Blood and lymphatic system disorders) | 11 (14) | 3 (5) | 7 (9)
Leukopenia (Blood and lymphatic system disorders) | 6 (27) | 0 (0) | 5 (13)
Lymphopenia (Blood and lymphatic system disorders) | 14 (26) | 2 (2) | 8 (21)
Neutropenia (Blood and lymphatic system disorders) | 12 (87) | 0 (0) | 7 (30)
Blepharitis (Eye disorders) | 4 (4) | 11 (16) | 0 (0)
Conjunctivitis (Eye disorders) | 4 (5) | 1 (1) | 1 (1)
Lacrimation increased (Eye disorders) | 4 (5) | 4 (4) | 4 (4)
Vision blurred (Eye disorders) | 1 (1) | 5 (6) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 5 (11) | 5 (5) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 6 (9) | 11 (20) | 6 (6)
Constipation (Gastrointestinal disorders) | 10 (14) | 7 (9) | 8 (10)
Diarrhoea (Gastrointestinal disorders) | 29 (65) | 29 (70) | 8 (10)
Dyspepsia (Gastrointestinal disorders) | 5 (6) | 7 (11) | 5 (6)
Mouth ulceration (Gastrointestinal disorders) | 4 (8) | 6 (8) | 1 (1)
Nausea (Gastrointestinal disorders) | 21 (40) | 10 (11) | 17 (24)
Stomatitis (Gastrointestinal disorders) | 15 (49) | 9 (15) | 1 (1)
Vomiting (Gastrointestinal disorders) | 25 (37) | 10 (11) | 12 (14)
Asthenia (General disorders) | 12 (16) | 6 (7) | 6 (22)
Chest pain (General disorders) | 4 (4) | 12 (12) | 3 (3)
Fatigue (General disorders) | 20 (33) | 9 (11) | 17 (24)
Mucosal inflammation (General disorders) | 14 (27) | 7 (8) | 3 (5)
Oedema (General disorders) | 3 (3) | 1 (1) | 4 (4)
Oedema peripheral (General disorders) | 8 (24) | 1 (1) | 6 (7)
Pyrexia (General disorders) | 11 (21) | 3 (4) | 9 (14)
Herpes zoster (Infections and infestations) | 5 (5) | 1 (1) | 2 (2)
Paronychia (Infections and infestations) | 7 (11) | 14 (16) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 7 (10) | 4 (8) | 3 (3)
Urinary tract infection (Infections and infestations) | 4 (5) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 13 (19) | 1 (1) | 8 (9)
Aspartate aminotransferase increased (Investigations) | 12 (19) | 3 (5) | 7 (8)
Creatinine renal clearance decreased (Investigations) | 0 (0) | 1 (1) | 6 (7)
Haemoglobin decreased (Investigations) | 10 (21) | 4 (13) | 5 (7)
Neutrophil count decreased (Investigations) | 16 (70) | 1 (9) | 7 (21)
Platelet count decreased (Investigations) | 6 (11) | 0 (0) | 5 (20)
Weight decreased (Investigations) | 4 (5) | 7 (7) | 5 (6)
White blood cell count decreased (Investigations) | 16 (77) | 2 (15) | 8 (17)
Decreased appetite (Metabolism and nutrition disorders) | 23 (39) | 15 (24) | 19 (31)
Hyperglycaemia (Metabolism and nutrition disorders) | 8 (9) | 4 (4) | 7 (10)
Hyponatraemia (Metabolism and nutrition disorders) | 5 (7) | 4 (5) | 6 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (7) | 3 (3) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 8 (9) | 9 (9)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (7) | 3 (5) | 3 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (6) | 5 (8) | 4 (4)
Dizziness (Nervous system disorders) | 10 (12) | 2 (2) | 5 (5)
Headache (Nervous system disorders) | 14 (16) | 8 (11) | 5 (5)
Paraesthesia (Nervous system disorders) | 4 (4) | 0 (0) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (4) | 0 (0) | 5 (5)
Insomnia (Psychiatric disorders) | 10 (18) | 10 (14) | 5 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 15 (18) | 28 (32) | 13 (17)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 (12) | 10 (10) | 10 (10)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 8 (11) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 1 (2) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 5 (7) | 6 (7) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 13 (21) | 2 (2)
Acne (Skin and subcutaneous tissue disorders) | 6 (10) | 3 (3) | 1 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 9 (9) | 2 (2) | 2 (4)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 10 (19) | 5 (5) | 1 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 12 (15) | 25 (26) | 2 (2)
Nail disorder (Skin and subcutaneous tissue disorders) | 3 (3) | 6 (6) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 17 (25) | 20 (35) | 4 (5)
Rash (Skin and subcutaneous tissue disorders) | 41 (57) | 43 (52) | 8 (14)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 5 (5) | 12 (14) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days